CLINICAL TRIAL: NCT04204694
Title: Study of the Role of Interferon αon the Endothelial Dysfunction During Septic Shock
Acronym: INTERSEP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7350
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient in septic shock
  Interventions: Other: 3-time blood sampling for septic shock patients
- blood donor tests
  Interventions: Other: Only one blood sampling for controls patients

INTERVENTIONS:
Other: 3-time blood sampling for septic shock patients — 15 mL blood are sampled at day1, day 3 and day 7, from the arterial catheter inserted for all patients with septic shock
  Groups: Patient in septic shock
Other: Only one blood sampling for controls patients — 15 mL blood are sampled from a blood donation
  Groups: blood donor tests

SUMMARY:
Septic shock is the most severe form of a bacterial infection, affecting 24 million patients per year worldwide, with a high mortality (> 30%).

Septic shock is defined by an acute circulatory failure, with low blood pressure and insufficient oxygen supply to organs. This circulatory failure is related to vascular damages, in which the endothelial vascular tissue is impaired by inflammatory mechanisms, with release of circulating endothelial cells in the blood.

Therefore, modulating inflammation on the vascular endothelial tissue could be a therapeutic strategy, and the investigators focus on the role of the type I interferons on the endothelial tissue because of the demonstrated role of type I interferons during septic shock.

Thus the investigators proceed to an observational study, in which the primary purpose will be to show a higher expression of type I interferon receptors on circulating endothelial cells in patients with septic shock compared to control subjects.

Concerning secondary purposes, the investigators will record mortality at d3, d7 and d28, perform assays about types I, II and III interferons in plasma, and test anti-interferon on endothelial cells ex vivo

ELIGIBILITY:
* For all subjects
* Age > 18 years old
* For females: negative pregnancy test
* Subject covered by health insurance
* Written consent
* Patients with septic shock
* Patients must be in ICU
* Septic shock defined by the Sepsis-3 criteria [1]
* Inclusion within the 12 hours following the onset of norepinephrin
* Controls :
* Blood donors

Exclusion criteria:

* Moribund
* Age < 18 years old
* Absence of written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will have two groups :
  1. Patients with septic shock hospitalized in the ICU from Strasbourg University Hospital
  2. Controls: blood donors recruited by the French blood establishment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Expression of the activated interferon-α receptors (IFNAR) by circulant endothelial cells | Within 12 hours following the onset of norepinephrin for septic shock (day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de réanimation médicale, Strasbourg, France